CLINICAL TRIAL: NCT02736084
Title: A Positive Psychology Program for Patients With Type 2 Diabetes: A Pilot Study
Brief Title: Boosting Emotions & Happiness in Outpatients Living With Diabetes
Acronym: BEHOLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Attending Psychiatrist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013P001602
Record Dates: First submitted 2016-03-30; First posted 2016-04-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Type 2 Diabetes
Keywords: optimism; positive affect; adherence; health behavior; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Health Behavior; Diabetes Mellitus | interventions — Psychology, Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Positive Psychology (Experimental): The Positive Psychology intervention consists of 7 exercises that will be completed by the participant with the guidance of a trainer.
  Exercises:
  Gratitude for positive events Using personal strengths Gratitude letter Enjoyable and meaningful activities Recalling past success Performing acts of kindness Repeating one of the previous exercises.
  Interventions: Behavioral: Positive Psychology

INTERVENTIONS:
Behavioral: Positive Psychology — The Positive Psychology intervention consists of 7 exercises that will be completed by the participant with the guidance of a trainer.

SUMMARY:
The investigators developed a novel, telephone-based, 12-week positive psychology intervention and will assess its feasibility and short-term impact in adults with type 2 diabetes (T2D) and suboptimal health behavior adherence. Participants will receive a positive psychology (PP) manual, complete exercises (e.g., writing a gratitude letter, performing acts of kindness), and review these activities by phone with a study trainer over the 12-week study period.

Specific Aim #1 (Feasibility and acceptability (immediate impact); primary aim): To assess whether PP exercises administered over the phone are feasible and linked with immediate benefit in patients with T2D, as measured by ratings provided pre- and post- each exercise.

Hypothesis: The PP exercises will be feasible (i.e., 4 of the 7 PP exercises will be completed by a majority of participants, and participants will have a mean score of at least 7 out of 10 on ratings of ease of completion for the exercises. The PP exercises will also have adequate immediate impact (i.e., mean ratings of 7/10 of exercise utility post-exercise and ratings of optimism post-exercise that are significantly higher than pre-exercise).

Specific Aim #2 (Changes in clinical outcome measures): To determine whether the PP intervention is linked to improvements in psychological well-being, during and after the intervention period (6 & 12 weeks), via measures of optimism, gratitude, depression, and anxiety. To examine whether the brief PP intervention is associated with improvements in self-reported outcomes related to health (diabetes self-care, diabetes distress, health related quality of life), during and after the intervention.

Hypothesis: Participants will have higher mean scores on all psychological outcome measures at 6 and 12 weeks compared to baseline. Participants will also have higher mean scores on all health-related outcome measures at 6 and 12 weeks compared to baseline.

DETAILED DESCRIPTION:
This is a pilot and feasibility study in adult inpatients and outpatients at MGH. Participants will have Type 2 Diabetes (T2D) and are required to report suboptimal adherence to health behaviors, measured by the Medical Outcomes Study Specific Adherence Scale (MOS SAS). All participants will receive a 12-week PP intervention and pre- and post-intervention assessments of mood and physical symptoms.

Participants will be enrolled from the outpatient Diabetes Center and inpatient medical units of MGH; research staff will introduce the study, assess for inclusion and exclusion criteria, and obtain written informed consent. Post-enrollment, and prior to initiation of the intervention, participants will complete baseline self-report measures of clinical outcomes.

During the initial enrollment visit, participants will receive a treatment manual. In person or by telephone, the study interventionist will review the introductory portion of the manual and discuss the first exercise (Gratitude for Positive Events) with the participant. In subsequent weeks, exercises will be completed independently by participants, recorded in their treatment manual, and then discussed over the phone with their trainer. In the final week, after the final exercise is reviewed, the interventionist and participant will discuss future implementation and ways to incorporate the principles into daily life.

The 12-week intervention will consist of 7 distinct PP exercises, to be completed weekly for the first 4 weeks and then biweekly over the next 8 weeks.

For feasibility, interventionists will record rates of exercise completion at each participant phone session. For acceptability, participants will rate their optimism and positive affect on a 0-10 scale prior to completing the exercise and then immediately following the exercise. Additionally, participants will also rate the ease and overall utility of the exercise on a 0-10 scale after each exercise.

At baseline, 6 weeks, and 12 weeks, non-interventionist study staff obtained the following validated measures of study outcomes:

* Optimism = Life Orientation Test-Revised (LOT-R)
* Gratitude = Gratitude Questionnaire-6 (GQ-6)
* Anxiety and depression = Hospital Anxiety and Depression Scale (HADS)
* Diabetes-related distress = Diabetes Distress Scale (DDS)
* Health-related quality of life and function = Patient-Reported Outcomes Measurement Information System physical function scale (PROMIS-PF-10)
* Diabetes self-care behaviors = Summary of Diabetes Self-Care Activities Measure (SDSCA)
* Health behavior adherence = Medical Outcomes Study Specific Adherence Scale (MOS SAS)

ELIGIBILITY:
Inclusion Criteria:

* Current patient of the MGH Diabetes Center or inpatient on Ellison 9-11, White 8-11, Ellison 16, or Bigelow 11
* Diagnosis of type 2 Diabetes (confirmed via medical record and patient's treatment provider)
* Age 18 and older
* Able to read/write in English
* Suboptimal adherence, defined as a score of 15 or less on three Medical Outcomes Study Specific Adherence Scale (MOS SAS) items related to adherence to medications, diet, and exercise.

Exclusion Criteria:

* Cognitive disorder precluding informed consent or meaningful participation in the PP exercises, assessed using a six-item cognitive screen developed for research.
* Lack of telephone access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Intervention Feasibility | 10 Weeks
  Rate of intervention feasibility will be measured by the number of exercises completed by each participant. After the exercise, participants will rate the ease of the exercise on a 0-10 Likert scale. Feasibility will be defined as: 4 of the 7 PP exercises will be completed by a majority of patients and subjects will have a mean score of at least 3.5 out of 5 on ratings of ease of completion for the exercises.
Intervention Acceptability | 10 weeks
  To assess acceptability (and immediate impact), participants will rate their optimism and positive affect on a 0-10 Likert scale prior to completing the exercise and then immediately following the exercise. Adequate immediate impact will be defined as: mean ratings of 3.5/5 of exercise utility post-exercise and ratings of optimism post-exercise that are significantly higher than pre-exercise.

SECONDARY OUTCOMES:
Change in LOT-R Scores | Baseline, 6 weeks, and 12 weeks
  The Life Orientation Test-Revised (LOT-R) is a validated, six item, self-report measure of optimism.
Change in GQ-6 Scores | Baseline, 6 weeks, and 12 weeks
  The Gratitude Questionnaire 6 is a brief, validated six-item measure of dispositional gratitude.
Change in HADS Scores | Baseline, 6 weeks, and 12 weeks
  The Hospital Anxiety and Depression Scale is a validated 14-item measure designed for medically ill patients and has few somatic symptom items.
Change in DDS Scores | Baseline, 6 weeks, and 12 weeks
  The 17-item Diabetes Distress Scale is a validated scale for use specifically in patients with diabetes
Changes in PROMIS-PF-10 Scores | Baseline, 6 weeks, and 12 weeks
  The Patient-Reported Outcomes Measurement Information System physical function scale is an NIH-supported 10-item scale used to asses health-related quality of life and function
Changes in SDSCA Scores | Baseline, 6 weeks, and 12 weeks
  11 items from Summary of Diabetes Self-Care Activities Measure Diabetes are used to measure self-care behaviors. Behaviors measured will be diet, physical activity, blood sugar monitoring, and foot care.
Changes in MOS SAS Scores | Baseline, 6 weeks, and 12 weeks
  Three Medical Outcomes Study Specific Adherence Scale items assessing medication, diet, and exercise, will be measured individually and as a composite score.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff C Huffman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DuBois CM, Millstein RA, Celano CM, Wexler DJ, Huffman JC. Feasibility and Acceptability of a Positive Psychological Intervention for Patients With Type 2 Diabetes. Prim Care Companion CNS Disord. 2016 May 5;18(3):10.4088/PCC.15m01902. doi: 10.4088/PCC.15m01902. eCollection 2016. PMID 27733954